CLINICAL TRIAL: NCT03544008
Title: Multicenter Retrospective International Survey to Evaluate the Rate of AXIOS-related AEs in Endoscopic Transmural Drainage of Pancreatic Fluid Collections
Status: Completed | Type: Observational
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Other Study IDs: Axios AEs
Record Dates: First submitted 2018-05-21; First posted 2018-06-01 (Actual); Last update posted 2021-03-18 (Actual); Status verified 2021-03

CONDITIONS: Endoscopic Transmural Drainage of Pancreatic Fluid Collections

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: The use of AXIOS in Endoscopic transmural drainage

SUMMARY:
This is a retrospective study. Electronic chart review at respective centers will be the only database used. No patient contact or additional procedures will be conducted.

The main objectives are:

A) To evaluate the use of AXIOS in Endoscopic transmural drainage of Pancreatic fluid collections (PFC) in terms of clinical success and technical success.

B) To assess the rates, management, need for re-intervention, need for surgery, etiology and characteristics of Pancreatic fluid collections (PFC) on the occurrence of AXIOS- related related adverse events(AE).

DETAILED DESCRIPTION:
This is a retrospective study. Electronic chart review at respective centers will be the only database used. No patient contact or additional procedures will be conducted.

Data that will be recorded on review of electronic medical record database include:

I. Demographics (age, gender) II. Indication for procedure III. Diagnosis and findings including radiologic findings IV. Prior endoscopy treatments V. Type and number of stents used VI. Pancreatic fluid collection location and measurements VII. Procedure time VIII. Technical success IX. Clinical success X. Adverse events XI. Management of adverse events XII. Recurrence of pancreatic fluid collections XIII. Follow-up time

The above data will be collected and recorded in an excel sheet. The data collection will be completely de-identified and password protected. The file will be emailed using an institution email and encrypted. The password will be given in a separate email or by phone call.

Inclusion:

All patients undergoing endoscopic management of pancreatic fluid collections between January 2011 to June 2017

Exclusion:

Age under 18

We will enroll 100 record between January 2011 to June 2017.

Time for collecting data:

1 month for data collection and 3 weeks for data analysis.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing endoscopic management of pancreatic fluid collections between January 2011 to June 2017

Exclusion Criteria:

* Age under 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients undergoing endoscopic management of pancreatic fluid collections between January 2011 to June 2017
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2011-01 (Actual); Primary Completion 2020-12 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
The investigators will evaluate the use of AXIOS in Endoscopic transmural drainage of Pancreatic fluid collections (PFC) | 24 months

SECONDARY OUTCOMES:
The investigators will assess the rates, management, need for re-intervention, need for surgery, etiology and characteristics of Pancreatic fluid collections (PFC) on the occurrence of AXIOS- related related adverse events(AE). | 24 months

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fugazza A, Sethi A, Trindade AJ, Troncone E, Devlin J, Khashab MA, Vleggaar FP, Bogte A, Tarantino I, Deprez PH, Fabbri C, Aparicio JR, Fockens P, Voermans RP, Uwe W, Vanbiervliet G, Charachon A, Packey CD, Benias PC, El-Sherif Y, Paiji C, Ligresti D, Binda C, Martinez B, Correale L, Adler DG, Repici A, Anderloni A. International multicenter comprehensive analysis of adverse events associated with lumen-apposing metal stent placement for pancreatic fluid collection drainage. Gastrointest Endosc. 2020 Mar;91(3):574-583. doi: 10.1016/j.gie.2019.11.021. Epub 2019 Nov 20. PMID 31759037